CLINICAL TRIAL: NCT01892163
Title: A Multicentre Prospective Open-label Randomised Clinical Trial Comparing the Efficacy of Fixed Versus PRN Dosing of 700 μg Dexamethasone Posterior Segment Drug Delivery System (Ozurdex) in Patients With Refractory Diabetic Macular Oedema
Brief Title: Multicentre Randomised Clinical Trial Comparing Fixed vs Pro re Nata (PRN) Dosing of 700 μg Dexamethasone
Acronym: OZDRY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: The Royal Wolverhampton Hospitals NHS Trust (Other Government); Frimley Park Hospital NHS Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sobha Sivaprasad, Consultant, Moorfields Eye Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIVS1007
Record Dates: First submitted 2013-06-25; First posted 2013-07-04 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema, Ozurdex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ozurdex PRN dosing (Active Comparator): Ozurdex PRN dosing versus Ozurdex fixed dosing
  Interventions: Device: Ozurdex
- Ozurdex fixed dosing (Experimental)
  Interventions: Device: Ozurdex

INTERVENTIONS:
Device: Ozurdex — Dexamethasone implant (Ozurdex)
  Other Names: Dexamethasone

SUMMARY:
Multicentre randomized controlled trial to evaluate whether 5 monthly fixed dosing of 700 µg Dexamethasone Posterior Segment Drug Delivery System (Ozurdex) is as efficacious as Optical coherence tomography (OCT)-guided PRN dosing in patients with refractory diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex aged 18 years or over
2. Diagnosis of diabetes mellitus (type 1 or type 2).
3. Best corrected visual acuity in the study eye between ≥34 and ≤73 ETDRS letters at 1m at baseline attributable to diabetic macular edema (DME)
4. On clinical exam at baseline in the study eye, retinal thickening due to diabetic macular oedema involving the centre of the macula and OCT central subfield > 300 microns despite previous therapy.
5. Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs.
6. Ability to return for study visits
7. Visual acuity in fellow eye ≥ 2/60
8. Ability to give informed consent throughout the duration of the study

Main Exclusion Criteria:

1. Macular ischaemia
2. Macular oedema is considered to be due to a cause other than diabetic macular oedema.
3. Co-existent ocular disease
4. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular oedema or alter visual acuity during the course of the study.
5. A substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sobha Sivaprasad, FRCS, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing
Started | 50 | 50
Completed | 48 | 49
Not Completed | 2 | 1
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 25 | 45
  >=65 years | 30 | 25 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.8) | 63.8 (11.1) | 64.6 (10.5)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 34 | 40 | 74
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between Arms in the Change From Baseline in Best Corrected Visual Acuity at 12 Months
Time Frame: Baseline and 12 months
Population: Intention to treat analysis (available case)
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing
Number analyzed (Participants) | 48 | 49
ETDRS letters | 0 (13.0) | 0.53 (16.1)

2. Secondary Outcome: Difference Between Arms in Change From Baseline Composite Scores of the National Eye Institute Visual Function Questionnaire (VFQ-25).
Description: NEI VFQ 25 is a questionnaire intended to measure visual function and quality of life. It has 25 questions. The original response of each item are coded as per the NEI VFQ scoring system ranging from 0 (lowest) to 100 (highest).
  Composite score = (Score for each item with a non-missing answer) / Total number of items with non-missing answers 100 = Best, 0 = Worst possible score
Time Frame: Baseline and 12 months
Population: Though 48 patients completed the trial in the PRN arm, one patient did not complete the questionnaire completely, making it invalid for analysis. Hence the PRN arm number for this outcome was 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing
Number analyzed (Participants) | 47 | 49
units on a scale | -0.45 (12.2) | 3.02 (15.4)

3. Secondary Outcome: Difference Between Arms in Change in Central Subfield Thickness.
Description: Central subfield thickness is defined as the average thickness in the central 1mm diameter circle of the ETDRS grid and is measured in microns
Time Frame: Baseline and 12 months
Population: Few patients in both groups developed cataract. Due to the dense cataract, it was not possible to obtain the macular scans. Hence the discrepancy between the population who completed the study and the number for whom the OCT was obtained at exit visit.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing
Number analyzed (Participants) | 47 | 47
microns | -90.1 (96.2) | -179.9 (172.4)

4. Secondary Outcome: Proportion of Patients With Ocular and Systemic Serious Adverse Events
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing
Number analyzed (Participants) | 50 | 50
participants | 10 | 9

ADVERSE EVENTS:
Time Frame: 1 year (between baseline and exit)
Arm/Group | Ozurdex PRN Dosing | Ozurdex Fixed Dosing
Serious Adverse Events (participants affected / at risk) | 10/50 | 9/50
Other Adverse Events (participants affected / at risk) | 13/50 | 8/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex PRN Dosing (N=50) | Ozurdex Fixed Dosing (N=50)
Death (Vascular disorders) | 1 | 1
Retinal Detachment (Eye disorders) | 0 | 1
cataract surgery in study eye (Eye disorders) | 4 | 1
Endophthalmitis (Eye disorders) | 1 | 0
Other non specific eye problems (Eye disorders) | 1 | 1
other non ocular events (Cardiac disorders) | 3 (3) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex PRN Dosing (N=50) | Ozurdex Fixed Dosing (N=50)
Raised Intraocular Pressure (Eye disorders) | 13 (13) | 8 (8)
vitreous haemorrhage (Eye disorders) | 3 | 3
cataract progresion (Eye disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes